CLINICAL TRIAL: NCT01916915
Title: The Effect of Addition of Tramadol to Levobupivacaine in Continuous Wound Infusion for Postoperative Pain Treatment in Cesarean Section
Brief Title: Usage of Tramadol With Levobupivacaine for Pain Treatment After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Perihan Ekmekçi, Associate Professor, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/06
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tramadol 1 (Experimental): 1 mg/kg tramadol + 0.25% levobupivacaine 4 ml/h infusion
  Interventions: Drug: Tramadol infusion via wound catheter; Drug: Levobupivacaine
- Tramadol 2 (Experimental): 2mg/kg tramadol + 0.25% levobupivacaine 4 ml/h infusion
  Interventions: Drug: Tramadol infusion via wound catheter; Drug: Levobupivacaine
- Levobupivacaine (Placebo Comparator): 0.25% levobupivacaine 4ml/h infusion
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Tramadol infusion via wound catheter
  Arms: Tramadol 1; Tramadol 2
Drug: Levobupivacaine

SUMMARY:
Patients experience considerable amount of pain after cesarean section. The aim of this study is to investigate the effect of tramadol (an opioid pain killer) added to levobupivacaine (a local anesthetic) in continuous wound infusion (which is done by placing a catheter in the incision) after cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Planned cesarean section
* American Society of Anesthesiologists Class I-II

Exclusion Criteria:

* Patients refusing to enroll in the study
* Serious coagulopathy
* Serious systemic disease
* Story of allergy to drugs being used in the study
* Morbid obesity (Body mass index > 30)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
lowering of pain as measured by visual analogue scores | forty eight hours after the operation

SECONDARY OUTCOMES:
total additional analgesic consumption | forty eight hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Perihan Ekmekçi, Associate Professor, Principal Investigator — Ufuk University Dr Rıdvan Ege Hospital Department of Anesthesiology and Reanimation
Locations (1):
- Ufuk University Dr Rıdvan Ege Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No